CLINICAL TRIAL: NCT02079103
Title: Virtual Reality Based Training - a Motivating and Effective Way of Regaining Arm Motor Function After Stroke? The VIRTUES Trial: A Multi-center RCT
Brief Title: Virtual Reality Training for Upper Extremity After Stroke
Acronym: VIRTUES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Sunnaas Rehabilitation Hospital (Other); Regionshospitalet Hammel Neurocenter (Other); Regionshospitalet Viborg, Skive (Other); KU Leuven (Other); Jessa Hospital (Other); The Research Council of Norway (Other); Helse Vest (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Principal Investigator, Iris Ch. Brunner, PhD, PT, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UiB-228792
Record Dates: First submitted 2014-02-27; First posted 2014-03-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: Virtual reality; Stroke; Arm motor function; Neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual reality (Experimental): Virtual reality training using the YouGrabber® for patients with impaired arm motor function after stroke. The YouGrabber exercises focus on intensity, repetitions and motivating tasks and are adapted to the patient's motor abilities.
  Interventions: Device: Virtual Reality
- Conventional arm training (Active Comparator): The patients receive supervised self-training exercises with focus on functional tasks adapted to their motor abilities.
  Interventions: Behavioral: Conventional arm training

INTERVENTIONS:
Device: Virtual Reality — During a 4 weeks period the patients will be offered 4-5 Virtual reality training sessions weekly of 45-60 minutes duration in addition to other rehabilitation. The Virtual reality training will be supervised by a physical or an occupational therapist. Virtual reality gaming parameters are adapted according to improving arm motor function.
  Other Names: YouGrabber®
  Arms: Virtual reality
Behavioral: Conventional arm training — During a 4 weeks period the patients will be offered 4-5 supervised self-training sessions weekly of 45-60 minutes duration in addition to other rehabilitation. The training will be task-related and supervised by a physical or an occupational therapist. Exercises increase in difficulty according to improving arm motor function.
  Arms: Conventional arm training

SUMMARY:
Background: High intensity training of challenging tasks with many repetitions is a key factor for regaining motor function after stroke. Novel virtual reality (VR) rehabilitation systems provide the potential to increase intensity and offer challenging and motivating tasks. The efficacy of VR systems has not been demonstrated yet in sufficiently powered studies.

Methods: In 5 participating rehabilitation centers patients in the subacute phase after stroke will be randomized to either a group receiving 4 weeks of VR training in addition to conventional arm training or a group receiving dose-matched and therapist attention-matched conventional arm-training.

Hypothesis: VR training is more effective in improving arm motor function than conventional arm training in the subacute phase after stroke.

DETAILED DESCRIPTION:
Background: Approximately two thirds of patients with stroke experience impaired arm motor function, which compromises independence in activities of daily living, occupational areas and quality of life. High intensity training of challenging tasks with many repetitions are key factors for regaining motor function after stroke. Novel virtual reality (VR) rehabilitation systems provide the potential to increase intensity and offer challenging and motivating tasks. The efficacy of VR systems has not been demonstrated yet in sufficiently powered studies.

Methods: In this study 120 patients in 5 participating Norwegian, Danish and Belgian rehabilitation institutions will be randomized to either a group receiving VR training in addition to conventional arm training or a group receiving dose-matched and therapist attention-matched conventional arm-training. During a period of 4 weeks the patients will be offered additional 4-5 training sessions weekly of 45-60 minutes duration by a physiotherapist or an occupational therapist. Arm motor function, dexterity and independence in daily life activities will be evaluated at baseline, post and 3 months follow-up assessments with the Action Research Arm Test, Box and Blocks Test and the Functional Independence Measure. Patient satisfaction and therapist satisfaction with the implementation of a new technology based rehabilitation system will also be assessed with questionnaires and interviews.

Objective: The objective of the VIRTUES trial is to study the effectiveness and acceptance of a novel VR training approach. The study will provide evidence-based knowledge of new virtual reality based treatment strategies to clinicians, patients and health economists.

ELIGIBILITY:
Inclusion Criteria:

* First ever ischemic or hemorrhagic stroke or former stroke without any residual motor impairment
* 1 - 12 weeks post stroke
* Impaired arm motor function but some residual arm motor activity as defined by a score of less than 52 on Action Research Arm Test (ARAT), and the ability to execute at least 20 degrees of active shoulder extension and abduction against gravity.

Exclusion Criteria:

* Severe cognitive impairment defined as < 20 on Mini Mental Status Examination
* Orthopedic impairment, limiting mobility substantially or causing pain
* Visual disorders limiting the ability to comply with treatment regimen - < 18 years
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Action Research Arm Test score from baseline | Baseline, after 4 weeks and at 3 months follow-up
  Assessment of changes in arm motor function from baseline to 3 months follow up

SECONDARY OUTCOMES:
Change in Box and Blocks Test score from baseline | Baseline, after 4 weeks, and at 3 months follow-up
  Assessment of dexterity
Change in Functional Independence Measure from baseline | Baseline, after 4 weeks, and 3 months follow-up
  Assessment of independence in daily life activities
ABILHAND questionnaire | After 4 weeks of intervention and at 3 months follow-up
  Self-reported use of both hands in daily life activities

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sture Skouen, MD, PhD, Study Director — University of Bergen, Helse Vest; Iris Brunner, PhD, Principal Investigator — University of Bergen, Helse Vest
Locations (5):
- Rehabilitation Campus Sint-Ursula, Herk-de-Stad, Belgium
- Denmark (2):
  - Hammel Neurocenter, Hammel
  - Skive Neurorehabilitation, Skive
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Sunnaas Rehabilitation Hospital, Nesoddtangen

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Brunner I, Skouen JS, Hofstad H, Assmus J, Becker F, Sanders AM, Pallesen H, Qvist Kristensen L, Michielsen M, Thijs L, Verheyden G. Virtual Reality Training for Upper Extremity in Subacute Stroke (VIRTUES): A multicenter RCT. Neurology. 2017 Dec 12;89(24):2413-2421. doi: 10.1212/WNL.0000000000004744. Epub 2017 Nov 15. PMID 29142090
- [Derived] Brunner I, Skouen JS, Hofstad H, Assmuss J, Becker F, Pallesen H, Thijs L, Verheyden G. Is upper limb virtual reality training more intensive than conventional training for patients in the subacute phase after stroke? An analysis of treatment intensity and content. BMC Neurol. 2016 Nov 11;16(1):219. doi: 10.1186/s12883-016-0740-y. PMID 27835977
- [Derived] Brunner I, Skouen JS, Hofstad H, Strand LI, Becker F, Sanders AM, Pallesen H, Kristensen T, Michielsen M, Verheyden G. Virtual reality training for upper extremity in subacute stroke (VIRTUES): study protocol for a randomized controlled multicenter trial. BMC Neurol. 2014 Sep 28;14:186. doi: 10.1186/s12883-014-0186-z. PMID 25261187